CLINICAL TRIAL: NCT06341309
Title: Exploratory Study of Irinotecan Liposomes Combined With Bevacizumab in Maintenance Therapy of Metastatic Colorectal Cancer
Brief Title: Exploratory Study of Irinotecan Liposomes in Maintenance Therapy of Metastatic Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Meng Qiu, Dr, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DEY-CRC-K09
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — irinotecan sucrosofate; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- irinotecan liposome injection combined with bevacizumab (Experimental): Patients will be treated with irinotecan liposome injection combined with bevacizumab. Treatment until the disease progresses, intolerable toxicity occurs, and the patient withdraws informed consent (whichever comes first).
  Interventions: Drug: Irinotecan Liposome; Drug: Bevacizumab

INTERVENTIONS:
Drug: Irinotecan Liposome — 70 mg/m^2 , d1, 14 days per cycle. Until the disease progresses, intolerable toxicity occurs, and the patient withdraws informed consent (whichever comes first).
Drug: Bevacizumab — 5mg/kg, d1, 14 days per cycle. Until the disease progresses, intolerable toxicity occurs, and the patient withdraws informed consent (whichever comes first).

SUMMARY:
To evaluate the progression-free survival (PFS1), objective response rate (ORR), disease control rate (DCR), progression-free survival from first-line treatment initiation (PFS2), overall survival (OS), and safety of irinotecan liposome combined with bevacizumab in patients with advanced metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18~85 years old.
* Histopathologically confirmed patient with an inoperable metastatic colorectal adenocarcinoma.
* pMMR or MSS.
* CR, PR, or SD (according to RECIST v1.1 criteria) achieved after 12-16 weeks of intensive treatment with a first-line chemotherapy regimen containing irinotecan/fluorouracil or a three-drug chemotherapy regimen containing oxaliplatin/irinotecan/fluorouracil plus bevacizumab.
* If previously received neoadjuvant or adjuvant therapy, the time interval between initiation of systemic first-line therapy and the date of last dosing must be at least 6 months.
* ECOG 0~1, patients ≥75 years old need an ECOG score of 0.
* Normal bone marrow and organ function: ① Neutrophils (ANC) ≥1.5×10^9/L, platelets (PLT) ≥75×10^9/L, hemoglobin (Hb) ≥85g/L, albumin (ALB) ≥30 g/L, white blood cells (WBC) ≥3.0×10^9/L, and no bleeding tendency; ② AST, ALT and alkaline phosphatase (ALP) were all ≤2.5× upper limit of normal range (ULN), and ≤5×ULN when liver metastases occurred; The total bilirubin level doesn't exceed the upper limit of the agency's normal range; Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance ≥60 ml/min (calculated according to Cockroft-Gault).
* Understand the situation of this study, patients and/or legal representatives voluntarily agree to participate in this study and sign informed consent form.

Exclusion Criteria:

* Known or suspected central nervous system metastasis.
* Had received surgery or other treatment for tumors other than intensive treatment (including chemotherapy, radiotherapy, research treatment, etc., within 4 weeks prior to enrollment, if the interval between the current treatment was longer than 5 drug half-lives, could be included).
* Previous treatment-related toxicity did not return to NCI-CTCAE v5.0 I or below (except for alopecia, peripheral neuropathy).
* The use of CYP3A, CYP2C8, and UGT1A1 inhibitors or inducers couldn't be discontinued or were not discontinued within 2 weeks prior to enrollment.
* The presence of severe gastrointestinal dysfunction or gastrointestinal perforation, intraperitoneal abscess, and fistula.
* Intestinal obstruction, signs and symptoms of intestinal obstruction, or the stent has been previously implanted and the stent has not been removed before the screening period.
* Interstitial lung disease.
* Tendency of arterial embolism and massive bleeding within 6 months before enrollment (except surgical bleeding).
* Patients with fluid accumulation that couldn't reach a stable state but small amount of ascites on imaging without clinical symptoms could be enrolled.
* Any serious or uncontrolled systemic disease, including uncontrolled high blood pressure, heart disease, active bleeding, active viral infection, etc.
* Have had other malignancies within the past 5 years or currently, except cured cervical carcinoma in situ, uterine carcinoma in situ, and non-melanoma skin cancer.
* Patients of childbearing age who refuse to take contraceptives, women who are pregnant or breastfeeding.
* The researchers didn't consider it appropriate to participate in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-09 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival -1 | From initial medication to the date of first documented progression or end of medication, whichever came first . Assessed up to 18 months.
  The time from initiation of maintenance therapy to first recording of PD or death, whichever occurs first. To investigate antitumor efficacy of study.

SECONDARY OUTCOMES:
Progression free survival -2 | The time from the start of first-line treatment to the maintenance of PD treatment or death, whichever occurs first. Assessed up to 24 months.
  The time from the start of first-line treatment to the maintenance of PD treatment or death, whichever occurs first. To investigate antitumor efficacy of study.
Objective response rate | From initial medication to the date of first documented progression or end of medication, whichever came first. Assessed up to 18 months
  To investigate antitumor efficacy of study.
Disease control rate | From initial medication to the date of first documented progression or end of medication , assessed up to 18 months.
  To investigate the preliminary antitumor efficacy of study.
Overall survival | From initial medication to the date of death from any cause, Assessed up to 30 months.
  To investigate antitumor efficacy of study.
Incidence of adverse events and severity of adverse events as assessed by CTCAE 5.0 | Assessed up to 6 months.
  To assess the incidence and severity of adverse events in combination regimens.